CLINICAL TRIAL: NCT00103584
Title: A Phase I/II Clinical Trial to Evaluate the Safety and Immunogenicity of LC16m8, A Modified Vaccinia Vaccine, in Healthy Volunteers
Brief Title: Safety and Immunogenicity Study of LC16m8, a Modified Smallpox Vaccine, in Healthy, Previously Unvaccinated Volunteers
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: VaxGen (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VAX012
Record Dates: First submitted 2005-02-10; First posted 2005-02-11 (Estimated); Last update posted 2007-01-15 (Estimated); Status verified 2007-01

CONDITIONS: Smallpox
MeSH Terms: conditions — Smallpox | interventions — smallpox vaccine LC16m8

INTERVENTIONS:
Biological: LC16m8 Smallpox Vaccine

SUMMARY:
This is a Phase I/II study evaluating the safety and immunogenicity of LC16m8, a modified vaccinia vaccine. After consent and thorough screening (including safety labs, EKG, and medical history), healthy, previously unvaccinated volunteers between the ages of 18-34 will receive a single vaccination of either LC16m8 or the current US-licensed smallpox vaccine, Dryvax. Volunteers will be blindly randomized to a treatment group in a 4:1 ratio (4 LC16m8 to 1 Dryvax recipient). Follow-up clinical evaluations, laboratory testing, EKGs and cardiac assessments will be done at regularly scheduled follow-up visits for 1 year after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the study and give written informed consent. A signed informed consent must be in place prior to any study procedures being performed.
* Male or female aged 18-34 years old (inclusive; year of birth = 1971-1987).
* No history of smallpox vaccination or evidence of vaccine site scar.
* Willing and able to return for all follow-up visits, study procedures, and blood draws for the duration of the study.
* In good health, as ascertained by medical history, clinical assessment, and baseline (screening) laboratory assessments.
* Negative ELISA for HIV or, if indeterminate, Western blot or other assay confirming that the serostatus does not reflect HIV infection.
* Negative Hepatitis B Virus (HBV) and Hepatitis C Virus (HCV) serology.
* Negative urine glucose by urinalysis (UA).
* ALT <1.5 times upper limit of normal.
* Adequate renal function as defined by serum creatinine ≤1.5 mg/dL; urine protein <100 mg/dL, or trace or negative proteinuria by UA, and an estimated creatinine clearance of >55 mL/min. Renal function is measured to ensure that subjects could meet criteria for use of Vistide, should this be needed.
* Hematocrit, hemoglobin, platelets, and white blood cell count (WBC) within normal limits for males and females.
* EKG and EEG (for those being tested) baseline readings within normal limits (these will be read at a central site).
* Willing to refrain from donating blood (other than study-related) throughout the study and for a period of at least 21 days (or until scab separation) after vaccination. In some cases, state laws are more restrictive.
* Negative serum pregnancy test for females at screening and within 2 days prior to vaccination.
* If the volunteer is female and of childbearing potential, she must agree to use effective birth control methods and not become pregnant during the course of the study. A female is considered to have childbearing potential unless post-menopausal or surgically sterilized. Effective birth control methods include licensed, approved hormonal methods such as pills, patch, injection, or implant.

Exclusion Criteria:

* Planning to move within 52 weeks from the time of vaccination.
* Known allergy to any materials used in this study or components of the vaccines, which may include erythromycin, streptomycin, chlortetracycline, polymyxin B, neomycin, phenol, glycerin, Vaccinia Immune Globulin (VIG), immunoglobulin, blood products containing immunoglobulin preparations, cidofovir, probenecid, and/or bandage adhesive tape.
* Pregnant or breastfeeding, or have close contact** with someone who is pregnant or breastfeeding.
* Active or past history of atopic dermatitis or eczema, or close contact** with someone with active or past history of atopic dermatitis or eczema.
* Presence of (or close contact** or sharing a household with) a skin condition with extensive breaks in the skin such as burns, impetigo, contact dermatitis, or zoster (shingles) not likely to heal by the day of vaccination.
* Darier's disease or close contact** with Darier's disease.
* Immunosuppression (including HIV), or close contact** with an immunosuppressed individual.
* Using immunosuppressive medications, in eye drops, by mouth, or topically (corticosteroid nasal sprays and inhalers are permissible at low doses after discussion with VaxGen Medical Monitor).
* Close contact** with children under 1 year old.
* Active or past malignancy with the exception of non-metastatic skin cancers.
* History of exuberant keloid formation.*
* Known cardiac disease or three or more cardiac risk factors (high blood pressure, diabetes mellitus, smoking, hypercholesterolemia, heart disease at age 50 or earlier in a first-degree relative, or obesity [defined as Body Mass Index (BMI)>30]).
* Currently under treatment for high blood pressure.
* History of solid organ or bone marrow transplantation.
* Evidence of immunosuppression or autoimmune disease, cardiac disease, renal disease, splenectomy, or unstable medical condition as determined by baseline medical history, physical assessment, or laboratory assessments.
* Neurological or psychological condition that may place volunteer at heightened risk from vaccination.
* Psychiatric condition that precludes compliance with the protocol.
* Received or plan to receive live vaccines 30 days before or after study vaccination.
* Received or plan to receive subunit or killed vaccines 14 days before or after study vaccination.
* Received or plan to receive immunoglobulin or other blood products 60 days prior to HIV screening or study vaccination.
* Received or plan to receive experimental drugs/vaccines 30 days before study vaccination or prior to study completion.
* Received or plan to receive systemic immunosuppressive therapy or radiation therapy 30 days before study vaccination or prior to study completion.
* Served in military conflicts and received smallpox vaccination, or military service prior to 1989.

  * As determined by the Principal Investigator (PI).

    * Close contact = frequent physical contact or sharing linen/clothing.

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150
Dates: Start 2004-10; Study Completion 2006-07

PRIMARY OUTCOMES:
Safety and immunogenicity

CONTACTS AND LOCATIONS:
Overall Officials: Marc Gurwith, MD, JD, Study Director — VaxGen
Locations (4):
- United States (4):
  - Stanford University, General Clinical Research Center, Stanford, California
  - University of Kentucky, Kentucky Clinic, Lexington, Kentucky
  - St. Louis University, Center for Vaccine Development, St Louis, Missouri
  - Vanderbilt University Medical Center, General Clinical Research Center, Nashville, Tennessee

REFERENCES:
- [Derived] Kennedy JS, Gurwith M, Dekker CL, Frey SE, Edwards KM, Kenner J, Lock M, Empig C, Morikawa S, Saijo M, Yokote H, Karem K, Damon I, Perlroth M, Greenberg RN. Safety and immunogenicity of LC16m8, an attenuated smallpox vaccine in vaccinia-naive adults. J Infect Dis. 2011 Nov;204(9):1395-402. doi: 10.1093/infdis/jir527. Epub 2011 Sep 15. PMID 21921208